CLINICAL TRIAL: NCT06044064
Title: "Effect of Screening Using Imaging (CT/ EUS) on Early Detection of Pancreatic Ductal Adenocarcinoma (PDAC) in Patients With New Onset Diabetes (NOD)" - A Prospective Pilot Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: PDAC-NOD-001
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: interventions — CA-19-9 Antigen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: A blood sample for CA 19-9 (cancer detection test) — * A blood sample for CA 19-9 (cancer detection test) levels will be taken at baseline.
  * Contrast CT abdomen - Pancreas protocol will be done at baseline.
  * EUS (Endoscopic Ultrasound) under moderate sedation will be done at baseline to you.
  * If suspicious lesion is found on examination, Fine Needle Aspiration - FNA will be done.

SUMMARY:
To assess whether EUS (Endoscopic Ultrasound) can serve as a valuable diagnostic tool for identifying PDAC at an early stage in individuals who have recently been diagnosed with diabetes.

Purpose: To improve the rates of early detection of pancreatic cancer.

Pancreatic ductal adenocarcinoma (PDAC) is a type of cancer that starts in the pancreas, a gland located in your abdomen. It happens when some cells in the pancreas start growing abnormally and form a cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Patients diagnosed with diabetes based on FBS/ PPBS/ HbA1C
* Presence of atleast 1 FBS parameter measured in the past 6-18 months which was not > 125 mg/dl
* END-PDAC score > 2

Exclusion Criteria:

* Known or newly detected chronic pancreatitis
* Past history of pancreatic cancer
* History of steroid use
* Contraindications for EUS

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients coming to OP will be screened at AIG for the study criterias, those who are meeting them, shall be enrolled after consent. Patients will enrolled for 1 year and followed up for 3 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PDAC at 3 years | 3yrs

SECONDARY OUTCOMES:
• Incidence of PDAC at baseline • Incidence of resectable PDAC at baseline • Incidence of resectable PDAC at 3 years | baseline and 3yrs